CLINICAL TRIAL: NCT00354068
Title: A Phase I Study of Imatinib Mesylate in Combination With Temozolomide in Patients With Malignant Glioma
Brief Title: Imatinib Mesylate and Temozolomide in Treating Patients With Malignant Glioma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: Pro00004364; DUMC-5514-06-1R2; NOVARTIS-DUMC-5514-06-1R2; CDR0000483760 (Other: NCI)
Record Dates: First submitted 2006-07-19; First posted 2006-07-20 (Estimated); Last update posted 2013-03-28 (Estimated); Status verified 2013-03

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult anaplastic oligodendroglioma; adult giant cell glioblastoma; adult gliosarcoma; adult mixed glioma; adult anaplastic astrocytoma; recurrent adult brain tumor; adult glioblastoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Oligodendroglioma; Glioblastoma; Gliosarcoma; Glioma; Astrocytoma; Brain Neoplasms | interventions — Imatinib Mesylate; Temozolomide

INTERVENTIONS:
Drug: imatinib mesylate
Drug: temozolomide
Other: pharmacological study

SUMMARY:
RATIONALE: Imatinib mesylate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving imatinib mesylate together with temozolomide may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of imatinib mesylate when given together with temozolomide in treating patients with malignant glioma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose and dose-limiting toxicity, if attainable, of imatinib mesylate in combination with temozolomide in patients with malignant glioma.
* Characterize the safety and tolerability of imatinib mesylate, including acute and chronic toxicities, in these patients.
* Determine the effect of temozolomide on the pharmacokinetics (PK) of imatinib mesylate at each dose level.
* Evaluate the impact of enzyme-inducing anti-epileptic drug (EIAED) coadministration on the PK of imatinib mesylate using a population-based PK approach.
* Evaluate the antitumor activity of imatinib mesylate plus temozolomide.

OUTLINE: This is a dose-escalation study of imatinib mesylate. Patients are stratified according to concurrent enzyme-inducing anticonvulsants (e.g., phenytoin, phenobarbital, carbamazepine, fosphenytoin, primidone, oxcarbazepine) (yes vs no).

Patients receive oral imatinib mesylate once or twice daily on days 1-8 and oral temozolomide once daily on days 4-8. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Cohorts of patients receive escalating doses of imatinib mesylate until the maximum tolerated dose is determined.

On days 1 and 8 of course 1, blood is drawn for pharmacokinetic studies.

PROJECTED ACCRUAL: A total of 40 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed malignant glioma

  * Any of the following subtypes:

    * Glioblastoma multiforme
    * Gliosarcoma
    * Anaplastic astrocytoma
    * Anaplastic oligodendroglioma
    * Anaplastic oligoastrocytoma
  * Previous histologic diagnosis of a lower grade of glioma allowed if there is histologic evidence of progression to a diagnosis of malignant glioma
  * Multifocal disease allowed
* Must have undergone prior conventional external-beam radiation therapy
* Stable disease, disease recurrence, or relapsed disease

  * Must not have received any systemic therapy for this recurrence or relapse
  * No prior progressive disease
* No central/systemic fluid collections (pericardial effusion, pulmonary effusion, ascites) ≥ grade 2
* No evidence of intratumor hemorrhage on pretreatment diagnostic imaging, except for stable post-operative grade 1 hemorrhage

PATIENT CHARACTERISTICS:

* Karnofsky performance status 70-100%
* Absolute neutrophil count > 1,500/mm³
* Hemoglobin > 9 g/dL
* Platelet count > 100,000/mm³
* AST and ALT < 2.5 times upper limit of normal (ULN)
* Bilirubin < 1.5 times ULN
* Creatinine < 1.5 times ULN
* No chronic renal disease
* No active uncontrolled infection
* No uncontrolled diabetes
* No excessive risk of bleeding, as defined by occurrence of any of the following:

  * Stroke within the past 6 months
  * History of CNS or intraocular bleed
  * Septic endocarditis
* No history of labile hypertension
* No congestive heart failure
* No poorly controlled hypertension
* No myocardial infarction within the past 6 months
* No history of poor compliance with antihypertensive regimen
* No other severe and/or uncontrolled medical disease that would preclude study participation
* No peripheral edema ≥ grade 2
* No gastrointestinal bleeding
* No gross hematuria
* No other active systemic bleeding
* Patients must not have experienced toxicity ≥ grade 3 with prior treatment with either temozolomide or imatinib mesylate
* No other primary malignancy within the past 5 years except basal cell skin cancer or carcinoma in situ of the cervix or other cancer not currently clinically significant nor requiring active interventions

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered from all prior therapy
* Prior surgical resection(s) allowed
* At least 2 weeks since prior surgery
* At least 2 weeks since prior chemotherapy (6 weeks for nitrosoureas)
* At least 2 weeks since prior external-beam radiotherapy
* At least 2 weeks since prior investigational drugs
* More than 1 week since prior biologic, immunotherapeutic, or cytostatic agents
* No concurrent warfarin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2004-07; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose
Dose-limiting toxicity
Safety and tolerability
Pharmacokinetics
Anti-tumor activity

CONTACTS AND LOCATIONS:
Overall Officials: David A. Reardon, MD, Study Chair — Duke Cancer Institute
Locations (1):
- Duke Cancer Institute, Durham, North Carolina, United States

REFERENCES:
- [Result] Reardon DA, Desjardins A, Vredenburgh JJ, Sathornsumetee S, Rich JN, Quinn JA, Lagattuta TF, Egorin MJ, Gururangan S, McLendon R, Herndon JE 2nd, Friedman AH, Salvado AJ, Friedman HS. Safety and pharmacokinetics of dose-intensive imatinib mesylate plus temozolomide: phase 1 trial in adults with malignant glioma. Neuro Oncol. 2008 Jun;10(3):330-40. doi: 10.1215/15228517-2008-003. Epub 2008 Mar 21. PMID 18359865